CLINICAL TRIAL: NCT05503771
Title: Health IT to Reduce Disparities in Risks for Sleep-related Infant Deaths, (SAFE Start 2.0 Project)
Brief Title: Improving Pediatrician Counseling About Infant Safe Sleep Using the Electronic Medical Record
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00333492; R01MD015818 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Sudden Infant Death; Sudden Unexplained Infant Death
Keywords: Counseling; Motivational Interviewing; Medical Informatics; Clinical Decision Support; Electronic Medical Record
MeSH Terms: conditions — Sudden Infant Death | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: ISA-MI (Experimental): The ISA-MI study condition involves, in addition to the standard of care described for the SOC group, a clinician training activity related to using the ISA (Infant Sleep Assessment) tool. Clinicians assigned to the ISA-MI Group will view a 20-30-minute recorded video training session on infant safe sleep (including its epidemiology, risk factors and recommendations), use of the ISA tool, and use of motivational interviewing-inspired (MI) communication skills to respond to ISA parent responses. The ISA tool builds on the 2022 AAP infant sleep recommendations and will be implemented at the 2-month WBV.
  Parents/patients of physicians in the ISA-MI study condition will also be given several infant safe sleep related products that facilitate compliance with safe sleep recommendations, namely, a portable crib, a sleep sack and a pacifier.
  Interventions: Behavioral: ISA-MI
- Control Group: Standard of Care (SOC) (Other): The SOC study condition consists of WBVs that follow the usual practice of American Academy of Pediatrics (AAP) Bright Futures Health Supervision Guidelines and includes age- and developmentally based anticipatory guidance. As part of their training, pediatric residents receive formal teaching on core aspects of providing primary care to infants, including the AAP recommendations on safe sleep. This includes the recommended ABCS: babies should sleep Alone (no objects or people), on their Back (supine), in a Crib (or safe alternative including portable crib or bassinet), and in a Smoke-free environment.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: ISA-MI — Parents seen by clinicians randomized to the intervention group will complete the Infant Sleep Assessment (ISA), either prior to their visit using MyChart (Epic patient portal) or on a tablet computer in the exam room while they wait for their clinician; 2) a Clinical Decision Support (CDS) smart form is created in the EMR based on the assessment results, with risks and MI-informed strategies highlighted; this information will be derived from a pre-programmed algorithm and theory-based, tailored communication strategies and messages; 3) the clinician uses the CDS smart form to guide counseling with the parent during the visit, applying their training in MI-informed counseling skills; and 4) Clinician gives the parent an After Visit Summary (AVS) from the EMR (or informs them that they can access the AVS in MyChart if the parent or other caregivers use the patient portal, MyChart), which summarizes and reinforces the safe sleep counseling.
  Arms: Intervention Group: ISA-MI
Other: Standard of Care (SOC) — Parents seen by clinicians randomized to the control group will receive the usual practice that pediatric residents are taught which follows the American Academy of Pediatrics (AAP) Bright Futures Health Supervision Guidelines and includes age and developmentally based anticipatory guidance. As part of their training, residents receive formal teaching on core aspects of providing primary care to infants, including the AAP recommendations on safe sleep. This includes the recommended ABCS: babies should sleep Alone (no objects or people), on their Back (supine), in a Crib (or safe alternative including portable crib or bassinet), and in a Smoke-free environment.
  Arms: Control Group: Standard of Care (SOC)

SUMMARY:
The study team will evaluate the impact of an Infant Sleep Assessment (ISA) tool with motivational interviewing (MI) communication training on clinician-parent communication during 2-month Well Baby Visits (WBV) and parent reported and observed infant sleep practices. The study team's hypotheses are that 1) clinicians who utilize the ISA with MI training will more effectively communicate safe sleep information to their patients' parents, and 2) these parents will have safer infant sleep practices than parents whose clinicians are in a standard of care control group.

DETAILED DESCRIPTION:
This research addresses the problem of unsafe infant sleep practices that increase the risk of Sudden Unexplained Infant Death (SUID), which includes Sudden Infant Death Syndrome and Accidental Suffocation and Strangulation in Bed. The study team will examine how a unique health information technology (HIT) tool impacts patient and provider outcomes when implemented in a pediatric primary care clinic serving a socioeconomically disadvantaged population that is primarily Black/African American. The study team's HIT tool - the Infant Sleep Assessment (ISA) - was developed through prior NIH-funded work and builds on the team's track record of innovative injury prevention research with parents and pediatric health care clinicians. During well-baby visits, the ISA assesses parents' reported sleep practices for their newborns. Using a programmed algorithm, the ISA identifies risky infant sleep practices and generates associated suggested feedback messages for the clinician that are derived from behavior change theory. This information is delivered via the electronic medical record (EMR) for the clinician's use during routine anticipatory guidance. To maximize the ISA's effectiveness, clinicians (pediatric residents) will receive a brief training in communication skills that are derived from Motivational Interviewing (MI). The study team will evaluate the impact of the ISA with MI communication training on clinician-parent communication during 2-month Well Baby Visits (WBV) and parent reported and observed infant sleep practices. The study team's hypotheses are that 1) clinicians who utilize the ISA with MI training will more effectively communicate safe sleep information to their patients' parents, and 2) these parents will have safer infant sleep practices than parents whose clinicians are in a standard of care control group.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish-speaking parents and legal guardians bringing their infants to the Harriet Lane Clinic (pediatric primary care clinic) for any of their early well baby visits (between 3-5 days up to 4 weeks of age)
* Maryland recognizes teen parents as emancipated minors, so they will be eligible to provide consent and participate.

Exclusion Criteria:

* Infant is considered medically complex (e.g., serious congenital anomaly, requires cardiorespiratory monitoring, etc.)
* Assigned resident is not enrolled in the study

Ages: 3 Days to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of infant safe sleep counseling provided by clinicians using new EMR-based tool as assessed by listening to recorded 2-month Well Baby Visits for control and intervention groups. | 2-month Well Baby Visit
  To test the impact of implementing a new EMR-based Infant Sleep Assessment (ISA) on pediatric clinicians' delivery of anticipatory guidance (both positive and unintended negative consequences) after watching a self-paced video training on safe sleep information, ISA tutorial, and motivational interviewing
Changes in quality of infant safe sleep counseling provided by clinicians trained in Motivational Interviewing skills as assessed by listening to recorded 2-month Well Baby Visits for control and intervention groups. | 2-month Well Baby Visit
  To test the impact of implementing a new EMR-based Infant Sleep Assessment (ISA) and brief Motivational Interviewing training (ISA-MI) on pediatric clinicians' delivery of anticipatory guidance (both positive and unintended negative consequences) after watching a self-paced video training on safe sleep information, ISA tutorial, and motivational interviewing
Changes in parents' satisfaction with care provided by clinical residents as assessed by the follow-up survey parents in both control and intervention groups will receive at the 4-month Well Baby Visit. | 4 months
  Asses parents' satisfaction with care, infant safe sleep knowledge, beliefs, reported practices, and observed infant sleep environments.

SECONDARY OUTCOMES:
Analyze clinicians' experiences with the ISA intervention as assessed by the clinician close-out survey when clinicians graduate or the study ends (whichever happens first). | Through Study Completion, an average of 2-3 years
  Assess clinicians' experiences with the ISA intervention, specifically reactions to using the ISA tool (preparation, satisfaction, ease of use, self-efficacy, burnout, impact on balancing measures).
Analyze ISA's advantages and disadvantages over standard anticipatory guidance as assessed by the clinician close-out survey when clinicians graduate or the study ends (whichever happens first). | Through Study Completion, an average of 2-3 years
  Assess clinicians' experiences with the ISA intervention, including: a) reactions to using the ISA (preparation, satisfaction, ease of use, self-efficacy, burnout, impact on balancing measures).
Review parents' experiences using the ISA tool as assessed by the Visit Exit Checklist (VEC) survey after the 4-month Well Baby Visit. | 4 months
  Perceptions of parents' reactions in the intervention group to using the ISA tool through MyChart.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Solomon, MD, MPH, Principal Investigator — Division of General Pediatrics; Eileen M McDonald, MS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Marisabel Cordon Villa de Leon, MPH, Study Director — Division of General Pediatrics
Locations (1):
- Harriet Lane Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No